CLINICAL TRIAL: NCT03374813
Title: Efficacy of MimetikOss in Alveolar Ridge Preservation Previous to Implant Placement: A Multicenter Randomized Controlled Trial.
Brief Title: Efficacy of MimetikOss in Alveolar Ridge Preservation Previous to Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mimetis Biomaterials S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REST-ECL-2017-01
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Alveolar Ridge Preservation
Keywords: Bone graft substitutes; Synthetic graft; Xenograft; Ridge preservation; Alveolar defect

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MimetikOss (Experimental): Ridge preservation bone grafting after tooth extraction
  Interventions: Device: MimetikOss (bone grafting surgery)
- Bio-Oss (Active Comparator): Ridge preservation bone grafting after tooth extraction
  Interventions: Device: Bio-Oss (bone grafting surgery)

INTERVENTIONS:
Device: MimetikOss (bone grafting surgery) — Ridge preservation bone grafting after dental extraction.
  Arms: MimetikOss
Device: Bio-Oss (bone grafting surgery) — Ridge preservation bone grafting after dental extraction.
  Arms: Bio-Oss

SUMMARY:
The hypothesis tested in this clinical trial is that a biomimetic synthetic bone graft substitute (MimetikOss, Mimetis Biomaterials) with similar properties to those of human bone can reach a clinical outcome non inferior to that of a deproteinized bovine bone matrix bone graft substitute (Bio-Oss, Geistlisch) in an alveolar ridge preservation procedure followed by implant placement in terms of bone volume changes (primary end point), bone histological observation implant stability and bone level changes (secondary end points).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old.
* Able to sign an informed consent form.
* Patients in need of socket preservation presenting 4 wall defects on premolar and molar zone in the maxilla or in the mandible.
* Healthy extraction site (no infected walls).
* The height of root molar bone support must be > 6 mm. The height of root molar bone support plus the bone height between the most apical root part and the sinus floor must be > 3 mm. As described in the picture below. Molar roots must be surgically separated previous to extraction
* Only 4 walled defects are included (3mm max of difference between buccal and lingual plate height).
* Presence of opposite occlusal dentition with natural roots in the area intended for extraction and implant placement.
* Natural roots are adjacent to implant site.
* If patient presents more than 1 defect that could be included in the study, only one will be part of the study, the other sites will be treated with the standard of care.
* Patient in good physical health.
* The subject is willing and able to comply with all study-related procedures (such as exercising oral hygiene and attending all follow-up procedures).
* Full-mouth bleeding score (FMBS) lower than 25%.
* The subject is suitable for a 2-stage surgical procedure.

Exclusion Criteria:

* Patients with premolar extraction due to the root fracture that present infected two wall type defect.
* Patients presenting the defect in the molar and/or premolar region of the maxilla with the concomitant need of sinus lift.
* Absence of adjacent teeth.
* Lack of opposite occluding dentition in the area intended for extraction and subsequent implant placement.
* 3 wall (or less) defects.
* Presence of bone dehiscence superior to 3 mm.
* Fenestration in the area intended to treat.
* Prior bone augmentation in the area planned for treatment (i.e ridge preservation).
* History of systemic diseases that would contraindicate oral surgical treatment or any other disease or medication that might have an influence on the involved tissues, such as intake of bisphosphonates, treatment with heparine, osteogenesis imperfecta, osteoporosis etc.
* Autoimmune disease (Rheumatoid polyarthritis, Crohn, Lupus, Sarcoidosis etc).
* Health conditions, which do not permit the surgical (including anaesthesia) or restorative procedure.
* Pregnant or breast feeding women.
* Any disorders directly in the planned implant area such as previous tumours, radiation or chronic bone disease.
* More than three teeth with full crown coverage in the dental arch (mandible or maxilla of the implant to be placed).
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, Paclitaxel, methotrexate etc).
* Active periodontal disease involving the residual dentition.
* Alcohol or drug abuse as noted in subject records or in subject history.
* Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or history.
* Heavy smoking (> 10 cigarettes per day).
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake or A1c level above 6.8%.
* Poor compliance.
* Mucosal diseases in the areas to be treated.
* Subject is involved in other clinical trial.
* Subject suffer severe bruxism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-04-22 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Bone volume changes | 6 months post grafting procedure
  Bone ridge horizontal and vertical change assessment by CBCT

SECONDARY OUTCOMES:
Bone histological observation | 6 months post grafting procedure
  Histomorphometric analysis of the tissue components
Implant survival | 4 months y 1 year post grafting procedure
  ISQ measurement and bone level changes analysis
Implant survival | 4 months y 1 year post grafting procedure
  Bone level changes analysis

CONTACTS AND LOCATIONS:
Locations (8):
- Universidad de los Andes, Santiago, Chile
- Spain (7):
  - IOC Dental Clinic, Vecindario, Las Palmas de Gran Canaria
  - Universitat Internacional de Catalunya, Barcelona
  - Universidad de granada, Granada
  - Clinica dental Triana, Las Palmas de Gran Canaria
  - Clínica Bustillo, Pamplona
  - Universitat de Sevilla, Facultad de odontología, Seville
  - Universidad de Valencia, Facultad de Medicina y Odontología, Valencia

IPD SHARING:
Plan to Share IPD: Undecided